CLINICAL TRIAL: NCT02374996
Title: Pharmacoepigenetics of Second Generation Antipsychotic-Induced Insulin Resistance in Bipolar Disorder
Brief Title: Pharmacoepigenetics of Bipolar Disorder Treatment
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Kyle Burghardt, Assistant Professor, Wayne State University
Other Study IDs: BPBIOPWSU
Record Dates: First submitted 2015-02-09; First posted 2015-03-02 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Antipsychotic Agents; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- APIGT: Bipolar subjects treated with antipsychotics and having impaired glucose tolerance
- APNGT: Bipolar subjects treated with antipsychotics and having normal glucose tolerance
- LINGT: Bipolar subjects treated with lithium and having normal glucose tolerance

SUMMARY:
Insulin is a hormone produced by the body to regulate blood sugar. Insulin resistance is a state when the body is not using insulin correctly, and more insulin is needed to maintain normal blood sugar. Insulin resistance is common in bipolar patients and even more common in bipolar patients treated with antipsychotics. Insulin resistance from antipsychotics can lead to type 2 diabetes, metabolic syndrome and cardiovascular disease and is known to lead to worse psychiatric outcomes (less mood stability) and lower life expectancies in bipolar disorder. Abnormal regulation of the folate cycle is known to play a role in antipsychotic-induced insulin resistance and the main endpoint to the folate cycle is the production of methyl donors for DNA methylation. DNA methylation is critical as it regulates how genes are expressed. Thus, changes in DNA methylation may play a role in the disease process of antipsychotic-induced insulin resistance. The purpose of this study is to examine the differences in the DNA methylation of candidate tissues known to have a role in the development of insulin resistance. The three groups of bipolar patients to be studied are 1) antipsychotic treated patients with impaired glucose tolerance, 2) antipsychotic treated patients with normal glucose tolerance and 3) lithium treated patients with normal glucose tolerance. Group 1 will be compared to groups 2 and 3 in order to assess how DNA methylation in the skeletal muscle and fat tissue changes due to medication effects (group 2 vs. 3) and medication side effects (group 1 vs. 2). Secondary analyses include the analysis of how fats are processed in skeletal muscle and fat tissue in relation to antipsychotic-induced insulin resistance and the correlation of DNA methylation across different tissues. The investigators hypothesize that antipsychotic-induced insulin resistance is to due changes in the way DNA is expressed (through epigenetic changes) which causes further changes in the way fats are processed in the body eventually leading to insulin resistance. This work is based on preliminary findings however further work is needed to identify the true mechanisms behind antipsychotic-induced insulin resistance and in particular, the main tissue in which this mechanism occurs.

DETAILED DESCRIPTION:
This study will be composed of 2 visits. The first visit will be used as a screening visit for inclusion of the three groups of patients for the second visit where the outcomes will be collected (e.g., tissue samples for DNA methylation and lipidomic analysis).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 with a Bipolar Spectrum Diagnosis (Bipolar I, II or NOS)
2. Currently treated with lithium or an antipsychotic as determined by a physician for at least 3 months at a stable dosage.
3. Non- obese with BMI < 30
4. Able to communicate meaningfully with the investigator and legally competent to provide informed written consent.
5. Females must be non-lactating, have a pregnancy test and be on acceptable birth control

105 subjects will be studied in total from three groups:

1. One group will consist of 35 bipolar patients currently stable on an antipsychotics with impaired glucose tolerance (2-hour postprandial plasma glucose of 140-199mg/dL).
2. The second group will consist of 35 age, gender, and body composition matched bipolar patients currently stable on an antipsychotic with normal glucose tolerance (2-hour postprandial plasma glucose <140mg/dL.
3. The third group will consist of 35 age, gender and body composition matched bipolar subjects stable on lithium with normal glucose tolerance.

Exclusion Criteria:

1. Currently diagnosed with diabetes (type I or II) or receiving treatment for diabetes. Any history of metabolic complications (weight gain, high cholesterol, high blood pressure) before taking an antipsychotic.
2. Active diagnosis of alcohol or substance abuse.
3. Primary relative diagnosed with type II diabetes.
4. Treated with any of the following medications: a) Systemic glucocorticoids (more than 2 weeks), antineoplastic agents, transplant medications, anti-retroviral medications within 6 months prior to screening.

   * Start or change of hormonal replacement therapy within 3 months prior to screening.
5. History or presence of any of the following conditions

   * Clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG)
   * Peripheral vascular disease (history of claudication)
   * Clinically significant pulmonary disease.
   * Current uncontrolled hypertension (systolic BP>160 mmHg, diastolic BP>100 mmHg)
   * History or presence of malignancy other than basal cell or squamous cell skin cancer
   * Clinically significant hematologic disease
6. Any of the following abnormal laboratory values:

   * Hematocrit < 35 vol%
   * Serum creatinine > 1.6 mg/dl
   * aspartate aminotransferase (AST), alanine aminotransferase (ALT) or Alkaline phosphatase > 2.5 times the upper limit of normal
   * Prothrombin time (PT), Partial thromboplastin time (PTT) outside the normal reference range
   * thyroid-stimulating hormone (TSH) outside the normal reference range
   * Triglycerides > 400 mg/dl
   * Platelet count < 50,000
7. Blood donation within 2 months prior to screening
8. Engage in exercise with moderate to hard intensity for greater than 1 hour per day for 5 or more days per week.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bipolar patients treated with Lithium or an antipsychotic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
DNA methylation in skeletal muscle and adipose tissue | Baseline
  The prevalence of DNA methylation of cytosine-phosphate-guanosine (CpG) Island 81 of the Fatty Acyl Coenzyme A Reductase gene will be compared amongst the groups. The is reported as % methylation

SECONDARY OUTCOMES:
shotgun Lipidomics in skeletal muscle and adipose tissue | Baseline
  shotgun lipidomics will be ran via the a lipidomics core in both muscle and adipose tissue. The quantified lipid metabolites (over 1000 will be quantified) will compared amongst groups using multivariate analyses

OTHER OUTCOMES:
DNA methylation Across tissues | Baseline
  Measure the correlation of DNA methylation in the fatty acyl coa reductase gene correlation across tissues (muscle vs. adipose vs. buccal)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle J Burghardt, PharmD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University Clinical Research Center, Detroit, Michigan, United States